CLINICAL TRIAL: NCT05650476
Title: Pre-approval Single-patient Expanded Access for Talazoparib (PF-06944076)
Status: Available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C344; NCT05650476 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Prostate Cancer; metastatic* Castration-Resistant Prostate Cancer (mCRPC); enzalutamide; combination therapy; first-line mCRPC; metastatic (M1)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — talazoparib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Talazoparib — capsules

SUMMARY:
Provide pre-approval single-patient Expanded Access (Compassionate Use) of talazoparib for patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
In Expanded Access, treating physicians are the Sponsors..

Expanded Access requests from treating physicians may be submitted at www.pfizercares.com; availability will depend on location/country.

ELIGIBILITY:
Talazoparib is not intended for monotherapy. Talazoparib is intended for combination use with enzalutamide in first-line metastatic (M1) Castration-Resistant Prostate Cancer (mCRPC) only. Must be a newly diagnosed mCRPC patient who has not yet received 1st line therapy (1st generation Androgen Receptor (AR)-inhibitors do not count). Must have not received 2nd generation AR-inhibitors (enzalutamide, apalutamide, darolutamide), a Poly [ADP-ribose] polymerase (PARP)-inhibitor, cyclophosphamide, or mitoxantrone as prior treatments in any prostate cancer disease setting. Previous abiraterone and/or docetaxel for hormone-sensitive disease (CSPC) is allowed (patient eligible). Patients with identified need for use of potent P-glycoprotein (P-gp) inducer drugs within 7 days of onset/under duration of talazoparib plus enzalutamide treatment are at risk of drug-drug interactions (DDIs) and are therefore ineligible. Additional eligibility criteria may be required.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult